CLINICAL TRIAL: NCT01220453
Title: Compliance and Efficacy in the Use of PICOPREP® for Bowel Cleansing
Brief Title: Compliance and Efficacy in the Use of PICOPREP®
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999169 CS01
Record Dates: First submitted 2010-10-05; First posted 2010-10-14 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Bowel Cleanliness

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The present trial is aimed to document efficacy (bowel cleanliness), acceptance and tolerability as well as patient comfort in the use of the new bowel cleansing product PICOPREP® in every day practice. In particular, it should be evaluated, whether bowel cleanliness, acceptance, tolerability and patient comfort are affected by specific practice procedures, changes in dose etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving PICOPREP® for bowel evacuation prior to endoscopy or surgery
* Patients who have been informed about the NIS and have given their written consent for participation

Exclusion Criteria:

* Patients in which prescription of PICOPREP® is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 2165 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Documentation of the use of PICOPREP® in every day practice | 2 days
  Will evaluate efficacy (bowel cleanliness), compliance, acceptance, tolerability and patient comfort

SECONDARY OUTCOMES:
Documentation of patient satisfaction after bowel cleansing | 2 days
Documentation of examiner satisfaction after colonoscopy | 2 days
Identification of patient groups in which bowel cleansing is more difficult due to concomitant diseases or other conditions (risk groups) | 2 days
Tolerability: frequency and severity of adverse events | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (121):
- Germany (121):
  - Investigational Site, Altdorf
  - Investigational Site, Altenholz
  - Investigational Site, Augsburg
  - Investigational Site, Bad Lausick
  - Investigational Site, Bad Schwalbach
  - Investigational Site, Bayreuth
  - Investigational Site, Beckum
  - Investigational Site, Berlin
  - Investigational Site, Bielefeld
  - Investigational Site, Bietigheim
  - Private Practice, Bietigheim-Bissingen
  - Investigational Site, Bitterfeld-Wolfen
  - Investigational Site, Bonn
  - Investigational Site, Brandenburg
  - Investigational Site, Braunschweig
  - Investigational Site, Brinkum
  - Investigational Site, Buchholz
  - Investigational Site, Butzbach
  - Investigational Site, Castrop-Rauxel
  - Investigational Site, Cologne
  - Investigational Site, Cottbus
  - Investigational Site, Dachau
  - Investigational Site, Detmold
  - Investigational Site, Dingolfing
  - Investigational Site, Dippoldswalde
  - Investigational Site, Dortmund
  - Investigational Site, Dresden
  - Investigational Site, Düsseldorf
  - Investigational Site, Eberswalde
  - Investigational Site, Elsterwerda
  - Investigational Site, Erftstadt
  - Investigational Site, Erfurt
  - Investigational Site, Eschweiler
  - Investigational Site, Essen
  - Investigational Site, Forchheim
  - Investigational Site, Frankfurt
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Friedrichshafen
  - Investigational Site, Gelsenkirchen
  - Investigational Site, Germering
  - Investigational Site, Giessen
  - Investigational Site, Giffhorn-Winkel
  - Investigational Site, Gilching
  - Investigational Site, Goslar
  - Investigational Site, Göppingen
  - Investigational Site, Grevenbroich
  - Investigational Site, Hagen
  - Investigational Site, Halle
  - Investigational Site, Haltern am See
  - Investigational Site, Hamburg
  - Investigational Site, Hamelin
  - Investigational Site, Hanover
  - Investigational Site, Haßloch
  - Investigational Site, Hebel
  - Investigational site, Hechingen
  - Investigational Site, Heinsberg
  - Investigational Site, Herne
  - Investigational Site, Herten
  - Investigational Site, Herzogenrath
  - Investigational Site, Hildesheim
  - Investigational Site, Hürth
  - Investigational Site, Itzehoe
  - Investigational Site, Jena
  - Investigational Site, Jerichow
  - Investigational Site, Juehlich
  - Investigational Site, Karlsruhe
  - Investigational Site, Karlstadt am Main
  - Investigational Site, Kassel
  - Investigational Site, Kiel
  - Investigational Site, Kitzingen
  - Investigational Site, Koblenz
  - Investigational Site, Königstein
  - Investigational Site, Königswusterhausen
  - Investigational Site, Landshut
  - Investigational Site, Leipzig
  - Investigational Site, Leverkusen
  - Investigational Site, Ludwigshafen
  - Investigational Site, Lübeck
  - Investigational Site, Magdeburg
  - Investigational Site, Mainz
  - Investigational Site, Mannheim
  - Investigational Site, Mönchengladbach
  - Investigational Site, Muenzenberg-Gambach
  - Investigational Site, München
  - Investigational Site, Münster
  - Investigational Site, Neubrandenburg
  - Investigational Site, Neumarkt
  - Investigational Site, Neumünster
  - Investigational Site, Neustadt
  - Investigational Site, Nienburg
  - Investigational Site, Nuremberg
  - Investigational Site, Oldenburg
  - Investigational Site, Paderborn
  - Investigational Site, Papenburg
  - Investigational Site, Plauen
  - Investigational Site, Polheim
  - Investigational Site, Potsdam
  - Investigational Site, Rheda
  - Investigational Site, Rinteln
  - Investigational Site, Rosenheim
  - Investigational Site, Rostock
  - Investigational Site, Rottach-Weissach
  - Investigational Site, Rottenburg
  - Investigational Site, Schwäbisch Hall
  - Investigational Site, Schweinfurt
  - Investigational Site, Siegen
  - Investigational site, Singen
  - Investigational Site, Stade
  - Investigational Site, Steinfurt
  - Investigational Site, Stuttgart
  - Investigational Site, Traunstein
  - Investigational Site, Uelzen
  - Investigational Site, Varel
  - Investigational Site, Waltrop
  - Investigational Site, Weißenburg
  - Investigational Site, Wertheim am Main
  - Investigational Site, Wesseling
  - Investigational Site, Wetzlar
  - Investigational Site, Wilhelmshaven
  - Investigational Site, Wittenberg
  - Investigational Site, Wriezen